CLINICAL TRIAL: NCT04264182
Title: STandardized Ultra-conservative Or Physician-directed ICD Programming for SHOCK Reduction Among Patients on Continuous Flow LVAD Support: a Randomized Controlled Trial (STOP SHOCK LVAD Study)
Brief Title: STandardized Ultra-conservative Or Physician-directed ICD Programming for Continuous Flow LVAD Support
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult to enroll patients into the study
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Dan Cantillon, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-656
Record Dates: First submitted 2020-01-31; First posted 2020-02-11 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Heart Failure, Systolic; Left Ventricular Assist Device; ICD
Keywords: LVAD; ICD; Shock; Ventricular arrhythmia
MeSH Terms: conditions — Heart Failure, Systolic; Shock

STUDY DESIGN:
Intervention Model Description: Prospective. Randomized control trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultra-conservative ICD programming (Experimental): Single VF zone programming strategy with maximal detection extension to avoid ICD shock delivery with monitoring-only VT detection zones
  Interventions: Other: ICD programming
- Standard programming (physician discretion) (No Intervention): Usual care ICD programming, which is historically unchanged from ICD programming pre-LVAD

INTERVENTIONS:
Other: ICD programming — Re-programming of the ICD device for VA detection (see above)
  Arms: Ultra-conservative ICD programming

SUMMARY:
This study will evaluate the utilization of an ultra-conservative programming strategy to reduce shocks for ventricular arrhythmias (VA) among patients with heart failure, an implantable cardioverter-defibrillator (ICD) and continuous flow (CF) left ventricular assist device (LVAD). Patients on LVAD support demonstrate unique hemodynamic tolerability of VA, and the role for ICDs among patients with newer generation CF LVADs remains less clear than the older generation devices. Prior studies have explored extended detection ICD programming to reduce unecessary or potentially avoidable shocks to patients. However, no prospective randomized study to-date has evaluated such programming strategies in the CF LVAD patient population. The study hypothesis is that ultra-conservative (UC) ICD programming will result in a reduction of shocks and an improvement in quality of life without increasing hospitalizations, syncope or death among patients on CF LVAD support, and the primary design is a 1:1 randomization between UC programming over standard, physician discretion programming.

DETAILED DESCRIPTION:
The current International Society for Heart and Lung Transplantation (ISHLT) guidelines provide a class I recommendation for tachy-therapy re-activation in patients with ICDs undergoing LVAD implantation. However, these guidelines reflect a survival benefit observed in cohorts comprised primarily of older-generation pulsatile flow LVADs. While the overall VA prevalence in the LVAD population exceeds 50% with VA usually occurring >200 beats per minute, VA are generally well-tolerated both hemodynamically and symptomatically. Observed LVAD flows do decrease during sustained VA but there are multiple case reports of LVAD patients remaining awake and asymptomatic despite hours of ventricular fibrillation and a large case series reported no deaths and rare syncope due to VA in CF LVAD patients. Contrary to guidelines, contemporary evaluations restricted to CF LVADs show no clear ICD survival benefit in single center studies nor a large, pooled meta-analysis. In fact, propensity-matched analyses of CF LVAD patients in the INTERMACS and UNOS registries have demonstrated increased mortality and more hospitalizations among patients with an active ICD and treated VA. It is unclear in the CF LVAD population whether ICD shocks themselves are harmful or rather identify a higher-acuity patient subgroup. In the general HF population, however, shocks have consistently been associated with worse outcomes. Shock reduction programming resulted in reduced mortality in the MADIT-RIT trial, suggesting shocks may be directly harmful and not only a marker of substrate.

Therefore, the present study will evaluate whether ultra-conservative (UC) programming for ICDs can reduce shocks over standard (physician-discretion) programming among patients with heart failure on CF LVAD support. The model is 1:1 randomization between the two programming strategies for patients with newly implanted CF LVAD devices and a pre-existing ICD. They will be eligible for enrollment during their index hospitalization, and after discharge up to their first outpatient follow-up visit no later than 3 months post discharge. The primary endpoints will be any ICD shock, all-cause mortality, and syncope. The secondary endpoints will be time to first ICD shock, time to first ICD shock for VT/VF, quality of life questionnaire and hospitalizations, including for heart failure and ventricular arrhythmias. The principal exclusion criteria will be pediatric patients, or those without a functional ICD system. Standard of care follow-up will continue thru 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Pre-existing ICD
* LVAD placement

Exclusion Criteria:

* Non-functional ICD system
* Uncontrolled ventricular arrhythmias within 7 days of enrollment (defined as VT/VF >30 seconds and/or causing hemodynamic instability and/or symptoms of pre-syncope or syncope)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
ICD shock delivery | Up to 24 months
  Number of patients with ICD shock delivery
Mortality | Up to 24 Months
  Incidence of all-cause death
Syncope | Up to 24 Months
  Individual occurrence of loss of consciousness

SECONDARY OUTCOMES:
Time to first ICD shock | Up to 24 Months
  Interval of time from baseline to first appropriate/non-appropriate ICD shock
Time to first ICD shock for VT/VF (appropriate shock) | Up to 24 Months
  Interval of time from baseline to first ICD shock for VT/VF (appropriate shock)
Standard INTERMACS survey | Up to 24 Months
  Quality of life measured by INTERMACS survey scored from 1 to 7
Hospitalization | Up to 24 Months
  Individual occurrence of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cantillon, M. D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT04264182/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/82/NCT04264182/ICF_001.pdf